CLINICAL TRIAL: NCT06916377
Title: The Economics of Domestic Violence: Evidence From Bangladesh
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Grand Challenges Canada (Other); Weiss Foundation (Unknown); World Bank - Sexual Violence Research Initiative (SVRI) (Unknown); Fund for Innovation in Development (Unknown); USAID Development Innovation Ventures (Unknown); The Agency Fund, International Growth Centre (IGC) (Unknown); National Science Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2000026184
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Intimate Partner Violence (IPV); Intimate Partner Violence Prevention
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Treatment assignment was stratified at the union level, the smallest administrative rural unit. From the two districts combined, a total of 88 unions were selected using Probability Proportional to Size (PPS). Each union contained 5 clusters (villages), yielding a total of 440 clusters. In each village, investigators randomly sampled 20 married couples aged 18-65, yielding a total of 8,800 married couples.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Norms with Private Delivery (Experimental): Soap opera that challenges harmful norms that condone IPV, targeting the belief that violence is an acceptable way to assert control or maintain reputation Private Delivery Mode: Men watch the soap opera privately at home on handheld devices.
  Interventions: Behavioral: Edutainment Content: Norms Campaign
- Norms + Skills with Private Delivery (Experimental): Soap opera that builds on the norms campaign by adding CBT-based skills for stress management and non-violent conflict resolution Private Delivery Mode: Men watch the soap opera privately at home on handheld devices.
  Interventions: Behavioral: Edutainment Content: Norms Campaign; Behavioral: Cognitive Behavioral Therapy (CBT)-based skills
- Placebo with Private Delivery (Experimental): Soap opera that features unrelated content to serve as a control group, isolating the effects of norms and resiliency messaging.
  Private Delivery Mode: Men watch the soap opera privately at home on handheld devices.
  Interventions: Behavioral: Edutainment Content: Placebo Campaign
- Norms with Public Delivery (Experimental): Soap opera that challenges harmful norms that condone IPV, targeting the belief that violence is an acceptable way to assert control or maintain reputation Public Delivery Mode: Men watch the soap opera publicly through community screenings.
  Interventions: Behavioral: Edutainment Content: Norms Campaign
- Norms + Skills with Public Delivery (Experimental): Soap opera that builds on the norms campaign by adding CBT-based skills for stress management and non-violent conflict resolution Public Delivery Mode: Men watch the soap opera publicly through community screenings.
  Interventions: Behavioral: Edutainment Content: Norms Campaign; Behavioral: Cognitive Behavioral Therapy (CBT)-based skills
- Placebo with Public Delivery (Experimental): Soap opera that features unrelated content to serve as a control group, isolating the effects of norms and resiliency messaging.
  Public Delivery Mode: Men watch the soap opera publicly through community screenings.
  Interventions: Behavioral: Edutainment Content: Placebo Campaign
- Norms with Private Delivery and Cash-for-Work program (Experimental): Soap opera that challenges harmful norms that condone IPV, targeting the belief that violence is an acceptable way to assert control or maintain reputation Private Delivery Mode: Men watch the soap opera privately at home on handheld devices.
  Cash-for-Work: Small weekly payments for viewing and providing feedback on the media content.
  Interventions: Behavioral: Edutainment Content: Norms Campaign
- Norms + Skills with Private Delivery and Cash-for-Work program (Experimental): Soap opera that builds on the norms campaign by adding CBT-based skills for stress management and non-violent conflict resolution Private Delivery Mode: Men watch the soap opera privately at home on handheld devices.
  Cash-for-Work: Small weekly payments for viewing and providing feedback on the media content.
  Interventions: Behavioral: Edutainment Content: Norms Campaign; Behavioral: Cognitive Behavioral Therapy (CBT)-based skills
- Placebo with Private Delivery and Cash-for-Work program (Experimental): Soap opera that features unrelated content to serve as a control group, isolating the effects of norms and resiliency messaging.
  Private Delivery Mode: Men watch the soap opera privately at home on handheld devices.
  Cash-for-Work: Small weekly payments for viewing and providing feedback on the media content.
  Interventions: Behavioral: Edutainment Content: Placebo Campaign
- Norms with Public Delivery and Cash-for-Work program (Experimental): Soap opera that challenges harmful norms that condone IPV, targeting the belief that violence is an acceptable way to assert control or maintain reputation Public Delivery Mode: Men watch the soap opera publicly through community screenings.
  Cash-for-Work: Small weekly payments for viewing and providing feedback on the media content.
  Interventions: Behavioral: Edutainment Content: Norms Campaign
- Norms + Skills with Public Delivery and Cash-for-Work program (Experimental): Soap opera that builds on the norms campaign by adding CBT-based skills for stress management and non-violent conflict resolution Public Delivery Mode: Men watch the soap opera publicly through community screenings.
  Cash-for-Work: Small weekly payments for viewing and providing feedback on the media content.
  Interventions: Behavioral: Edutainment Content: Norms Campaign; Behavioral: Cognitive Behavioral Therapy (CBT)-based skills
- Placebo with Public Delivery and Cash-for-Work program (Experimental): Soap opera that features unrelated content to serve as a control group, isolating the effects of norms and resiliency messaging.
  Public Delivery Mode: Men watch the soap opera publicly through community screenings.
  Cash-for-Work: Small weekly payments for viewing and providing feedback on the media content.
  Interventions: Behavioral: Edutainment Content: Placebo Campaign

INTERVENTIONS:
Behavioral: Edutainment Content: Norms Campaign — Soap opera that challenges harmful norms that condone IPV, targeting the belief that violence is an acceptable way to assert control or maintain reputation.
  Arms: Norms + Skills with Private Delivery; Norms + Skills with Private Delivery and Cash-for-Work program; Norms + Skills with Public Delivery; Norms + Skills with Public Delivery and Cash-for-Work program; Norms with Private Delivery; Norms with Private Delivery and Cash-for-Work program; Norms with Public Delivery; Norms with Public Delivery and Cash-for-Work program
Behavioral: Cognitive Behavioral Therapy (CBT)-based skills — CBT-based skills for stress management and non-violent conflict resolution.
  Arms: Norms + Skills with Private Delivery; Norms + Skills with Private Delivery and Cash-for-Work program; Norms + Skills with Public Delivery; Norms + Skills with Public Delivery and Cash-for-Work program
Behavioral: Edutainment Content: Placebo Campaign — Soap opera that features unrelated non-violent content
  Arms: Placebo with Private Delivery; Placebo with Private Delivery and Cash-for-Work program; Placebo with Public Delivery; Placebo with Public Delivery and Cash-for-Work program

SUMMARY:
This project aims to test the scalability and cost-effectiveness of edutainment-soap operas designed to challenge harmful social norms and promote resilience-as a strategy to improve mental health and reduce intimate partner violence (IPV) in rural Bangladesh. Investigators will run a clustered randomized control trial in which villages will be randomized to one of three versions of the same soap opera: (i) Norms: Challenges harmful norms that condone IPV, targeting the belief that violence is an acceptable way to assert control or maintain reputation, (ii) Norms + Skills: builds on the norms campaign by adding CBT-based skills for stress management and non-violent conflict resolution, (iii) Placebo: No violence content. Investigators will evaluate the impact on attitudes towards IPV and IPV incidence.

DETAILED DESCRIPTION:
Study design features two layers of commuity-level randomization based on a 3x2 factorial design:

First Treatment Variation: Edutainment Content. Communities are randomized into one of three versions of the same soap opera:

1. Norms Campaign (176 communities): Challenges harmful norms that condone IPV, targeting the belief that violence is an acceptable way to assert control or maintain reputation.
2. Norms + Skills Campaign (176 communities): Builds on the norms campaign by adding CBT-based skills for stress management and non-violent conflict resolution.
3. Placebo Campaign (88 communities): Features unrelated content to serve as a control group, isolating the effects of norms and resiliency messaging.

This variation allows for assessing the impact of addressing harmful norms alone from the additional benefits of equipping men with practical coping skills. By comparing the Norms Campaign to the Norms + Skills Campaign, investigators test whether adding stress-coping skills yields additional reductions in IPV and related outcomes.

Second Treatment Variation: Delivery Modes. Fifty percent of communities in each treatment arm are randomized into one of two delivery modes:

1. Private Delivery: Men watch the soap opera privately at home on handheld devices.
2. Public Delivery: Men watch the soap opera publicly through community screenings.

Randomizing delivery modes enables investigators to assess whether men's responses to the intervention are driven by self-esteem concerns (private delivery) or reputation concerns (public delivery). This distinction provides critical insights into the mechanisms underlying IPV and informs the scalability of different delivery methods.

In addition to the community-level randomizations, 50 percent of men in each community are randomized into participation in a cash-for-work program. This individual-level randomization allows us to evaluate the role of economic strain in IPV outcomes, testing whether alleviating financial stress enhances the intervention's effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* married men and women over the legal age of majority in Bangladesh

Exclusion Criteria:

* No exclusion criteria were imposed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Husband (male) and wife (female) from each household
Enrollment: 440 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Demographic and Health Survey (DHS) to assess Acceptability of IPV | 1 month post intervention
  Standardized attitudinal questions from the Demographic and Health Survey (DHS), which capture whether violence is considered justified in specific situations to measure changes in husbands' personal attitudes towards IPV. Measured by the average score on a justification index across treatments. This index is a normalized index of how justified men think it is for a husband to use IPV.
Hypothetical vignettes to assess Acceptability of IPV | 1 month post intervention
  Hypothetical vignettes, where respondents evaluate the likely and socially acceptable behavior of a hypothetical husband whose wife transgressed a gender norm. These vignettes mitigate social desirability bias and improve the accuracy of responses on sensitive topics to measure changes in husbands' personal attitudes towards IPV. Measured by the average level of violence respondents across treatments believe hypothetical husband will and should assign if the hypothetical wife transgresses. The scale will be between 0 and 5.
Hypothetical vignettes to assess Perceptions about others' acceptability of IPV. | 1 month post intervention
  Husbands' perceptions about others' attitudes towards IPV were measured using the hypothetical vignettes. Respondents estimate the attitudes of the other surveyed men in their community using visual aids and stickers, each representing a different respondent.
  Hypothetical vignettes, where respondents evaluate the likely and socially acceptable behavior of a hypothetical husband whose wife transgressed a gender norm. These vignettes mitigate social desirability bias and improve the accuracy of responses on sensitive topics to measure changes in husbands' personal attitudes towards IPV. This will be measured by the average level of violence respondents across treatments believe other men in their community will assign if the hypothetical wife transgresses. The scale will be between 0 and 5.
Use of coping strategies to assess Men's resilience and mental health. | 1 month post intervention
  Men's coping and emotional self-regulation strategies are measured using an index constructed from responses provided by their wives. This index includes selected questions on men's approaches to conflict management from the Revised Conflict Tactics Scale, adapted items from the Bengali version of the Brief Resilient Coping Scale that capture spouses' perceptions of men's behavior, and measures of substance use. IPV-related questions are intentionally excluded, as these behaviors represent a distinct conceptual category measured separately. To simplify interpretation, the index is standardized relative to the control group by subtracting the control group's mean and dividing by its standard deviation. Consequently, the resulting index has a mean of zero and a standard deviation of one within the control group. Higher values of the index indicate more positive coping styles and better emotional regulation.
Patient Health Questionnaire-9 (PHQ-9) to assess Men's resilience and mental health. | 1 month post intervention
  Husbands' self-reported symptoms of depression measured using the PHQ-9 scale. PHQ-9 is a 9-item validated questionnaire used to screen for depression with a range of scores from 0-45. A cumulative score of ≥10 is considered positive with lower scores indicating no or mild anxiety.
Stressors and experiences to assess Men's resilience and mental health. | 1 month post intervention
  Husbands' open-ended responses on daily stressors and positive experiences to measure husbands' resilience and emotional well-being. A summary index with two subcomponents is developed. First, a sub-index of daily events using an adapted version of the Daily Hassles and Uplifts Scale that includes items relevant to our target population. Second, a sub-index that aggregates men's appraisal of stressors and is based on the 10-item version of the Perceived Stress Scale validated in Bangladesh. Each subcomponent is standardized to have a mean of zero and a standard deviation of one for the control group. The summary index is defined as the equally weighted average of these standardized sub-indexes, with signs oriented so that higher values consistently indicate more favorable outcomes (fewer stressors and/or lower perceived stress).
Biometric stress indicators to assess Men's resilience and mental health. | 1 month post intervention
  Biometric stress indicators, captured by Empatica E4 wristbands during sensitive survey modules, measuring physiological markers of emotional regulation and stress to measure husbands' resilience and emotional well-being. Specifically, electrodermal activity (EDA) data, expressed in microsiemens (μS), is used to analyze Skin Conductance Responses (SCRs). SCRs are quantified using a trough-to-peak (TTP) analysis, where the amplitude of each response is measured as the difference between the peak and the preceding trough within a defined time window. To identify event-related SCRs, a response window of 1 to 5 seconds following a stimulus is applied, with a minimum amplitude threshold of 0.01 μS to detect significant responses. The primary outcome variable is the sum of SCR amplitudes for significant responses. The average sum of SCR amplitudes across treatment groups is compared to assess differences in physiological stress responses.
Adapted version of the DHS to assess Prevalence and frequency of IPV. | 1 month post intervention
  An adapted version of the DHS, covering physical, psychological, financial, and sexual violence. To enhance privacy and reduce misreporting, women use visual response tools to answer these questions privately to measure women's experiences of IPV. Measured by the average of a standardized IPV index. This is a normalized index which captures the frequency (never, very few times, sometimes, or very often) of women's reported experiences of IPV in the past six months. Higher values indicate higher frequency of IPV.
Number of participants with IPV-related injuries to assess Prevalence and frequency of IPV. | 1 month post intervention
  Enumerators' reports of visible IPV-related injuries, such as bruises, documented using a standardized reporting protocol. Enumerators receive specialized training to identify and record signs of physical violence, with a focus on facial bruises and scratches, which remain visible even for veiled women to measure women's experiences of IPV.
Health assessments to assess Prevalence and frequency of IPV. | 1 month post intervention
  Health assessments by community health workers, who check for IPV-related injuries to measure women's experiences of IPV. Measured by the percentage of female respondents across treatments on whom community health workers identify IPV-related injuries.
Incidence of IPV to assess Prevalence and frequency of IPV. | Baseline and 6-12 months post intervention
  Women's self-reports of IPV through rolling phone surveys six to twelve months post-intervention.
  Measured by the average of a standardized IPV index. This is a normalized index which captures the frequency (never, very few times, sometimes, or very often) of women's reported experiences of IPV in the past six months.

SECONDARY OUTCOMES:
Respectable man scale to assess Men's self-esteem. | 1 month post intervention
  Husbands' reports of the likelihood that they are a "respectable man". Investigators constructed the respectable man scale using a combination of qualitative and quantitative methods. Husbands answer ten embedded questions throughout the survey that contribute to their respectable man score. At the end of the interview, investigators inform men that the top five scorers in the community are considered "respectable men," but we do not reveal their actual scores to them. Husbands indicate how confident they are that they rank among the top five in their community. Measured by the mean likelihood that men across treatments think they rank among the top five respectable men in their community. The scale will be between 0 and 100.
Perceived respectabillity to assess Men's reputation | 1 month post intervention
  Husbands' perceived probability that two randomly selected community members would consider them respectable, elicited using an identical ten-bean method. To reduce misreporting, husbands receive financial incentives based on the accuracy of their estimates. Measured by the mean likelihood that men across treatments think others rank them among the top five respectable men in their community. The scale will be between 0 and 100.
Cost-effectiveness of the edutainment campaigns assessed by Reduction to IPV exposure | 1 month post intervention
  Reduction in the number of women exposed to IPV or the intensity of IPV in the last six months per USD 1,000.
  Multiply the observed reduction in IPV (either in absolute prevalence or an intensity index) caused by each edutainment campaign by the total number of men assigned to that campaign. Investigators will calculate costs by summing both start-up and implementation costs. Start-up costs include intervention development (content production and pilot testing), adaptation (translation and cultural adjustments), and set-up (community engagement and facilitator training). Implementation costs include broadcasting and screening expenses, facilitator compensation, and routine monitoring and evaluation. Research-related expenditures will be excluded and only include costs related to activities expected at scale.
Cost-effectiveness of the edutainment campaigns assessed by benefit-to-cost ratio | 1 month post intervention
  Benefit-to-cost ratio calculated by dividing the estimated benefits from reduced IPV by the total costs of intervention delivery. To estimate the benefits of IPV reduction, investigators will use the treatment effects on income and a web-based cost benefit analysis tool developed by one of the Principal Investigators. This tool calculates the lifetime economic returns to increased income.
Cost-effectiveness of the edutainment campaigns assessed by benefit-to-cost ratio | 1 month post intervention
  Net present value calculated as the difference in discounted benefits and costs. To estimate the benefits of IPV reduction, investigators will use the treatment effects on income and a web-based cost-benefit analysis tool developed by one of the Principal Investigators. This tool calculates the lifetime economic returns to increased income. The unit of measure for NPV is 1000 USD.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Buchmann, PhD, Principal Investigator — Yale University
Locations (1):
- BRAC University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No